CLINICAL TRIAL: NCT06938594
Title: Working With Your Body in the Operating Room. The Case of Operating Room Nurses
Brief Title: Working With Your Body in the Operating Room. The Case of Operating Room Nurses (RCIBO)
Acronym: RCIBO
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0311 - RCIBO
Record Dates: First submitted 2025-02-10; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Nurses; Operating Rooms
Keywords: operating room nurses; opened bodies; surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The undocumented observation, repeatedly observed in the operating rooms, of discomfort, including fainting, among medical and paramedical novices working in contact with surgical breaches raises questions about the mechanisms put in place to cope with what seems initially unimaginable. Indeed, accounts in the social sciences show that the surgical opening of a living person is, in some ways, a transgressive act, forbidden outside the operating room. By spilling blood, it induces a 'symbolic disorder' described by Mary Douglas, that is contained through ritualized practices, predispositions towards objectification, and injunctions to control affects. The use of surgical drapes allows for the partial erasure of the person being operated on, who is no longer seen as a subject, but as an object of care - a dehumanized body or 'image-object' described by Amandine Klipfel. It is possible that ORNs are gradually adapting to negotiate the reconfiguration of bodies in the operating room, the transgression inherent in the surgical opening of a living person, and the personal resonance this may have for them. The investigator questions the specificities of their profession and their physical, emotional, and cognitive relationships following the initial shock of confronting open bodies. Is it possible to grow accustomed to or adapt to open bodies to the point of no longer experiencing difficulties related to what was once unthinkable? The investigator aims to understand what becomes of these initially unrepresentable experiences and roles ORNs have in redefining the bodies present - the processes of objectification and rehumanization of patients in the operating rooms. This doctoral study grasps the cognitive and imaginary constructions they experience in France and Canada.

ELIGIBILITY:
Inclusion Criteria:

* operating room nurses
* Student nurses and operating room nurses
* Supervisors
* Doctors, interns and externs
* Surgeons
* Midwives and midwifery students
* Hospital cleaning staff
* Nursing assistants
* Biomedical staff

Exclusion Criteria:

* People not involved in surgical operations
* People refusing to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Operating room nurses
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
References to emotions in interviews | From enrollment to the end of treatment at 1 year

SECONDARY OUTCOMES:
Identification of body postures, verbal and non-verbal communication, reactions and interactions of professionals during observations in the operating rooms | From enrollment to the end of treatment at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement